CLINICAL TRIAL: NCT01919268
Title: Effectiveness of the Addition of the Interferential Current to the Pilates Method in the Treatment of Patients With Chronic Nonspecific Low Back Pain: a Randomized Controlled Trial
Brief Title: Addition of the Interferential Current to the Pilates Method in the Treatment of Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Cristina Maria Nunes Cabral, Associate Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 18034113.7.0000.0064
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Nonspecific Low Back Pain
Keywords: Pilates-based exercises; Electrotherapy; Interferencial current
MeSH Terms: interventions — Electric Stimulation Therapy; Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrotherapy (Experimental): Combination of active interferential current with exercises of the Pilates method. Patients will receive 18 sessions of treatment over a period of 6 weeks (3 sessions/week). The exercises of the Pilates method will be individualized to each patient's needs (pragmatic treatment).
  Interventions: Device: Electrotherapy
- Pilates (Active Comparator): Combination of placebo interferential current with exercises of the Pilates method. Patients will receive 18 sessions of treatment over a period of six weeks (3 sessions/week). The exercises of the Pilates method will be individualized to each patient's needs (pragmatic treatment).
  Interventions: Device: Pilates

INTERVENTIONS:
Device: Electrotherapy — Combination of active interferential current with exercises of the Pilates method. Patients will receive 18 sessions of treatment over a period of 6 weeks (3 sessions/week). The exercises of Pilates method will be individualized to each patient's needs (pragmatic treatment).
  Arms: Electrotherapy
Device: Pilates — Combination of placebo interferential current with exercises of the Pilates method. Patients will receive 18 sessions of treatment over a period of 6 weeks (3 sessions/week). The exercises of the Pilates method will be individualized to each patient's needs (pragmatic treatment).
  Arms: Pilates

SUMMARY:
This study aims to evaluate the effectiveness of the addition of the interferential current to Pilates method exercises in the treatment of 148 patients with chronic nonspecific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary patients with chronic nonspecific low back pain longer than 12 weeks
* Pain greater than three points in Pain Numerical Rating Scale

Exclusion Criteria:

* Contra indications to physical exercise
* Serious spinal pathologies (e.g. tumors, fractures and inflammatory diseases)
* Nerve root compromise
* Pregnancy
* Infection and/or skin lesions at the site of the application of the interferential current
* Cancer
* Cardiac pacemaker
* Changes in sensitivity or allergy in the region of electrode placement
* Previous surgery on spine or physical therapy for chronic nonspecific low back pain in the last six months
* Previous experience with the Pilates method

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Disability | Six weeks after randomization
  Disability associated with low back pain will be measured by the 24-item Rolland Morris Disability Questionaire
Pressure pain threshold | Six weeks after randomization
  Pressure pain threshold will be evaluated using a pressure algometer
Pain intensity | Six weeks after randomization
  Pain intensity will be measured by an 11-point Pain Numerical Rating Scale

SECONDARY OUTCOMES:
Pain intensity | Six months after randomization
  Pain intensity will be measured by an 11-point Pain Numerical Rating Scale
Disability | Six months after randomization
  Disability associated with low back pain will be measured by the 24-item Rolland Morris Disability Questionaire
Global impression of recovery | Six weeks and six months after randomization
  Global impression of recovery will be measured by an 11-point Global Perceived Effect Scale
Specific disability | Six weeks and six months after randomization
  Specific disability will be evaluated by an 11-point Patient-specific Functional Scale
Kinesiophobia | Six weeks and six months after randomization
  Kinesiophobia will be evaluated by the Tampa Scale for Kinesiophobia

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy Outpatient Department, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Franco KM, Franco YD, Oliveira NB, Miyamoto GC, Santos MO, Liebano RE, Cabral CN. Is Interferential Current Before Pilates Exercises More Effective Than Placebo in Patients With Chronic Nonspecific Low Back Pain?: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Feb;98(2):320-328. doi: 10.1016/j.apmr.2016.08.485. Epub 2016 Oct 19. PMID 27771359
- [Derived] Franco YR, Liebano RE, Moura KF, de Oliveira NT, Miyamoto GC, Santos MO, Cabral CM. Efficacy of the addition of interferential current to Pilates method in patients with low back pain: a protocol of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Dec 10;15:420. doi: 10.1186/1471-2474-15-420. PMID 25492853